CLINICAL TRIAL: NCT05492539
Title: Incidence and Risk Factors for Developing Infections in Patients Colonized by Carbapenemase-producing Klebsiella Pneumoniae
Brief Title: Incidence and Risk Factors for Developing Infections in Patients Colonized by CP-KPC
Acronym: KPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MARINA VALINOTI, Principal Investigaror, Hospital Italiano de Buenos Aires
Other Study IDs: 3978
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Carbapenemase-Producing Enterobacteriaceae
Keywords: Health Care Associated Infections; Carbapenemase-Producing Enterobacteriaceae; colonization status; Risk Factors
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
The worldwide increase in the rate of infections due to multidrug-resistant bacteria is considered a major public health problem.

Infections caused by carbapenem-resistant Klebsiella pneumoniae (CR-KP) are associated with high morbidity and mortality. Mortality of up to 70% and, in survivors, a readmission rate of up to 72% within 90 days of discharge have been reported.

CR-KP infection is usually preceded by colonization. However, the incidence rate and risk factors for CR-KP infections among carriers is poorly understood.

Multiple studies have focused in risk factors to develop infections among carriers.

In order to identify patients at low risk of CR-KP bloodstream infections, Gianella et at developed a predictive score to stratify patients according to their risk for acquisition of CR-KP infections.

However, further studies are needed to validate these results, particularly in high-risk patients, such as haematological patients, solid organ trasplant recipients and patients admitted in ICU.

Italian Hospital is an acute tertiary care university teaching hospital with more than 45,000 admission-years, in Buenos Aires, Argentina, with a great proportion of haematological and solid organ transplant recipients, and patients with substantial comorbidities and immunosuppression.

With the aim of developing an adequate risk assessment for CR-KP infections among CR-KP carriers, we performed a retrospective cohort analysis, in a tertiary teaching hospital in Buenos Aires, Argentina.

The main purpose of our study is to describe the incidence of CR-KP infections among CRKP colonized patients, to demonstrate the risk factors for acquisition of CR-KP infections and to develop a clinical predictive score that could stratify patients to guide therapeutic decisions in CR-KP carriers, and avoid overuse of broad-spectrum therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients with a CR-KP positive rectal swab, hospitalized from 01/2014 to 01/2019

Exclusion Criteria:

* Unwillingness to participate

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) patients with a CR-KP positive rectal swab, hospitalized in an acute tertiary care university teaching hospital in Buenos Aires, Argentina
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
CRKP infections in CRKP colonized patients | through study completion, an average of 1 year
  the presence of a positive clinical culture of CR-KP, a documented physician diagnosis, and the initiation of targeted antimicrobial therapy.

SECONDARY OUTCOMES:
30 day all-cause mortality | through study completion, an average of 1 year
  30-day mortality rate starting from the date the relevant clinical culture was obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Valinoti, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Giannella M, Trecarichi EM, De Rosa FG, Del Bono V, Bassetti M, Lewis RE, Losito AR, Corcione S, Saffioti C, Bartoletti M, Maiuro G, Cardellino CS, Tedeschi S, Cauda R, Viscoli C, Viale P, Tumbarello M. Risk factors for carbapenem-resistant Klebsiella pneumoniae bloodstream infection among rectal carriers: a prospective observational multicentre study. Clin Microbiol Infect. 2014 Dec;20(12):1357-62. doi: 10.1111/1469-0691.12747. Epub 2014 Aug 11. PMID 24980276
- [Result] Gutierrez-Gutierrez B, Salamanca E, de Cueto M, Hsueh PR, Viale P, Pano-Pardo JR, Venditti M, Tumbarello M, Daikos G, Pintado V, Doi Y, Tuon FF, Karaiskos I, Machuca I, Schwaber MJ, Azap OK, Souli M, Roilides E, Pournaras S, Akova M, Perez F, Bermejo J, Oliver A, Almela M, Lowman W, Almirante B, Bonomo RA, Carmeli Y, Paterson DL, Pascual A, Rodriguez-Bano J; Investigators from the REIPI/ESGBIS/INCREMENT Group. A Predictive Model of Mortality in Patients With Bloodstream Infections due to Carbapenemase-Producing Enterobacteriaceae. Mayo Clin Proc. 2016 Oct;91(10):1362-1371. doi: 10.1016/j.mayocp.2016.06.024. PMID 27712635
- [Result] Ny P, Nieberg P, Wong-Beringer A. Impact of carbapenem resistance on epidemiology and outcomes of nonbacteremic Klebsiella pneumoniae infections. Am J Infect Control. 2015 Oct 1;43(10):1076-80. doi: 10.1016/j.ajic.2015.06.008. Epub 2015 Jul 17. PMID 26190386